CLINICAL TRIAL: NCT01812356
Title: Study of Cryomaze Procedure Using Nitrous Oxide Versus Argon Gas
Brief Title: The Concomitant Cryomaze Procedure Using Nitreous Oxide Cryoprobe: Comparison With Argon Based Cryoprobe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-11-088
Record Dates: First submitted 2013-03-08; First posted 2013-03-18 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2016-03

CONDITIONS: Atrial Fibrillation; Valve
Keywords: Atrial fibrillation; maze operation; cryoablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Argon gas probe (Experimental): Cryomaze procedure using Argon gas probe
  Interventions: Device: Cryomaze procedure using Argon
- Nitrous oxide probe (Active Comparator): Cryomaze procedure using Nitrous oxide probe
  Interventions: Device: Cryomaze procedure using Nitrous oxide

INTERVENTIONS:
Device: Cryomaze procedure using Nitrous oxide — Cryomaze procedure using Nitrous oxide
  Other Names: Atricure cryoprobe
  Arms: Nitrous oxide probe
Device: Cryomaze procedure using Argon — Cryomaze procedure using Argon
  Other Names: ATS medtronic probe
  Arms: Argon gas probe

SUMMARY:
The aim of this study is compare the surgical convenience and early and long-term outcomes of cryomaze procedure using nitrous oxide with using Argon gas.

The investigators will analyze the pathologic findings of atrial tissue after cryoablation using two probes and early and long-term outcomes with Holter monitoring. Atrial fibrillation burden 3 months and 1 year postoperatively and atrial activity will be checked.

DETAILED DESCRIPTION:
The investigators have used the Medtronic ATS cryoprobe (Argon based) since 2009 for cryomaze procedure for treatment of atrial fibrillation combined with valvular heart disease.

However, sometimes, it was inconvenient due to excess flexibility, wide lesion related to excess low temperature and time-consuming detachment from atrium after cryoablation. The investigators introduced Atricure cryoprobe (Nitreos Oxide based) in hope of overcoming these shortcomings of ATS probes last year.

Up to date, the investigators have been satisfactory in terms of the surgical convenience. On the other hand, we have the questionability of transmural lesion of Atricure probe because of the higher temperature of Atricure probe compared with ATS probe.

The aim of this study is compare the surgical convenience and early and long-term outcomes of cryomaze procedure using nitrous oxide with using Argon gas.

The investigators will analyze the pathologic findings of atrial tissue after cryoablation using two probes and early and long-term outcomes with Holter monitoring. Atrial fibrillation burden 3 months and 1 year postoperatively and atrial activity will be checked.

ELIGIBILITY:
Inclusion Criteria:

* requiring concomitant maze operation with valve surgery (persistent atrial fibrillation)
* between 18 and 75 years old

Exclusion Criteria:

* previous cardiac surgery
* Behcet disease
* Takayasu's arteritis
* Infective endocarditis
* Congenital heart disease
* left atrial size over 80mm
* moderate or greater functional tricuspid regurgitation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
recurrence of atrial fibrillation | one year
  Treatment failure

SECONDARY OUTCOMES:
Postoperative stroke | one year
  Thromboembolism
Atrial arrhythmia events | one year
  AF recurrence, the need for antiarrhythmic drugs for symptoms, permanent pacemaker insertion, and the need for cardioversion
Cardiac related death | one year
  Including sudden death
heart failure | one year
  heart failure requiring admission
Reoperation | one year
  reoperation due to heart problems
Intracranial hemorrhage | one year
  bleeding complication involving brain

CONTACTS AND LOCATIONS:
Overall Officials: Pyo Won Park, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No